CLINICAL TRIAL: NCT02419131
Title: Coalition to Alleviate PTSD: Randomized Clinical Trial of Cognitive-Behavior Therapy for Posttraumatic Headache
Brief Title: Cognitive-Behavior Therapy for Posttraumatic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC2014339H
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Post-traumatic Headache; PTSD
MeSH Terms: conditions — Post-Traumatic Headache; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral Headache Therapy (Experimental): A standard, manualized behavioral intervention for primary headache disorders
  Interventions: Behavioral: Behavioral Headache Therapy
- Cognitive Processing Therapy (Experimental): A gold-standard treatment for PTSD, called Cognitive Processing Therapy
  Interventions: Behavioral: Cognitive Processing Therapy
- Treatment as Usual (Active Comparator): Treatment as usual, receiving standard care for PTHA
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Behavioral Headache Therapy — A standard, manualized behavioral intervention for primary headache disorders
  Arms: Behavioral Headache Therapy
Behavioral: Cognitive Processing Therapy — A gold-standard treatment for PTSD, called Cognitive Processing Therapy
  Arms: Cognitive Processing Therapy
Behavioral: Treatment as Usual — Treatment as usual, receiving standard care for PTHA
  Arms: Treatment as Usual

SUMMARY:
The overall purpose of the study is to compare two talk therapies (Clinic-Based Cognitive Behavioral Therapy and Cognitive Processing Therapy-Cognitive Only) for the treatment of posttraumatic headache (PTHA) and co-morbid posttraumatic stress (PTS). The researchers hope to learn if a non-medication, cognitive-behavioral treatment can result in noticeable reductions in PTHA intensity/severity and frequency as well as PTS symptom severity.

DETAILED DESCRIPTION:
More than 100,000 military service members and veterans suffer from chronic headaches resulting from a traumatic brain injury (TBI) sustained during deployment. Although that population has seen a sharp increase in these posttraumatic headaches (PTHA), the condition is extraordinarily difficult to treat. There is very little evidence guiding its management.

Complicating things is the fact that those who have suffered a traumatic injury during deployment often have co-occurring symptoms of posttraumatic stress, which may worsen their headaches or make them more difficult to treat.

To better inform our understanding of how to help our suffering war veterans, we developed a study for the Consortium to Alleviate PTSD (CAP) addressing posttraumatic headache in war veterans with co-occurring symptoms of posttraumatic stress.

A key aim of the study will be to evaluate whether a leading psychological therapy for migraine headaches is effective with posttraumatic headaches. Investigators also seek to determine if treatment for PTHA likewise improves problems with PTSD, and whether treatment for PTSD simultaneously alleviates headaches.

To accomplish these aims, the study will have three arms, with participants placed randomly into one of three treatment conditions:

1. Treatment as usual (e.g., receiving standard care for PTHA through the South Texas Veterans Health Care System's Polytrauma Rehabilitation Center in San Antonio);
2. A gold standard, manualized cognitive-behavioral intervention for headache; or
3. A gold-standard treatment for PTSD, called Cognitive Processing Therapy.

ELIGIBILITY:
Inclusion Criteria:

* adult (ages 18 - 70 years old)
* U.S. military Veterans with military service during Operations Enduring Freedom (OEF), Iraqi Freedom (OIF), and New Dawn (OND)
* have sustained a traumatic head injury
* have been diagnosed or report symptoms consistent with chronic (> 3 months) posttraumatic headache attributed to a traumatic injury sustained as part of military service. We are focusing on chronic PTHA due to the very low likelihood of headache remission after 3 months, the disability associated with chronic PTHA, and the high prevalence of chronic versus acute PTHA in this Veteran population. A positive PTHA diagnosis will be indicated for individuals with de novo headache onset within 3 months of a concussion or exacerbation of pre-existing headache symptoms (increased frequency, duration, or intensity) within 3 months of traumatic injury. This is consistent with the existing ICHD-III criteria for PTHA inclusion will be based on either a pre-existing diagnosis of chronic PTHA documented in the Veteran's medical record by a PRC/PSC provider or a Neurologist (e.g., ICD-10 code G44.329) or through screening with one of our PRC/PSC co-PIs if the Veteran reports symptoms consistent with chronic PTHA but has never had it documented in her/his medical record.
* Participants taking headache medication with a stable pattern of use for the prior 6 week period (including no prescribed changes in medical regimen).
* Participants must have some posttraumatic stress (PTS) symptoms based on a cut-off score of at least 25 or above on the PTSD CheckList -Version (PCL-5), which all participants will complete as part of their screening.
* Participants must also report on the Clinician Administered PTSD Scale (CAPS-5) an exposure to a traumatic event (Criterion A), at least one intrusion symptom (Criterion B), and at least one avoidance symptom (Criterion C). There is some evidence suggesting 40% comorbidity between PTSD and new onset headache, so it is reasonable to assume that at least half of all PTHA participants recruited for this study will have PTHA and comorbid PTS symptoms. The inclusion of PTS symptoms in this sample is vital based on reports indicating that PTS symptoms and PTSD actually increase vulnerability to PTHA and chronic headache in military populations

Exclusion Criteria:

* there has been a recent and significant change in the nature of headache symptoms over the last 6 weeks prior to their screening (as determined by the investigators)
* Participants currently in CPT or prolonged exposure for PTSD.
* Participant has medication overuse headache as defined by the Structured Diagnostic Headache Interview-Revised (Brief Version; SDIHR).
* the participant is unable to read or speak English at a 6th grade level
* they have had a psychiatric hospitalization in the last 12 months
* they currently meet a psychiatric diagnosis of substance abuse [based on Alcohol Use Disorders Identification Test (AUDIT) assessment during screening]
* they are pregnant or plan to become pregnant during the trial (due to concerns about pregnancy-induced headache that may obscure findings)
* if a psychiatric problem is present that warrants immediate treatment based upon clinical judgment
* if they demonstrate significant cognitive impairment that could impact treatment adherence/benefit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald McGeary, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- San Antonio VA Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing as per CAP (Consortium to Alleviate PTSD) established protocol.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study completion when summary results are posted on ClinicalTrials.gov

REFERENCES:
- [Derived] McGeary DD, Resick PA, Penzien DB, McGeary CA, Houle TT, Eapen BC, Jaramillo CA, Nabity PS, Reed DE 2nd, Moring JC, Bira LM, Hansen HR, Young-McCaughan S, Cobos BA, Mintz J, Keane TM, Peterson AL. Cognitive Behavioral Therapy for Veterans With Comorbid Posttraumatic Headache and Posttraumatic Stress Disorder Symptoms: A Randomized Clinical Trial. JAMA Neurol. 2022 Aug 1;79(8):746-757. doi: 10.1001/jamaneurol.2022.1567. PMID 35759281
- [Derived] Moring JC, Straud CL, Penzien DB, Resick PA, Peterson AL, Jaramillo CA, Eapen BC, McGeary CA, Mintz J, Litz BT, Young-McCaughan S, Keane TM, McGeary DD. PTSD symptoms and tinnitus severity: An analysis of veterans with posttraumatic headaches. Health Psychol. 2022 Mar;41(3):178-183. doi: 10.1037/hea0001113. PMID 35298210
- [Derived] McGeary DD, Resick PA, Penzien DB, Eapen BC, Jaramillo C, McGeary CA, Nabity PS, Peterson AL, Young-McCaughan S, Keane TM, Reed D, Moring J, Sico JJ, Pangarkar SS, Houle TT; Consortium to Alleviate PTSD. Reason to doubt the ICHD-3 7-day inclusion criterion for mild TBI-related posttraumatic headache: A nested cohort study. Cephalalgia. 2020 Oct;40(11):1155-1167. doi: 10.1177/0333102420953109. Epub 2020 Aug 31. PMID 32867535

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who were consented and randomized, but did not continue to therapy
Period: Consent and Randomization
Arm/Group | Behavioral Headache Therapy | Cognitive Processing Therapy | Treatment as Usual
Started | 65 | 64 | 64
Completed | 55 | 48 | 57
Not Completed | 10 | 16 | 7
Not completed — Did not receive treatment after randomization | 10 | 16 | 7
Period: Randomization and Treatment
Arm/Group | Behavioral Headache Therapy | Cognitive Processing Therapy | Treatment as Usual
Started (Started treament) | 55 | 48 | 57
Completed 3-month Follow-up | 31 | 21 | 40
Completed 6-month Follow-up | 32 | 23 | 40
Completed Post-Treatment Follow-up | 33 | 23 | 48
Completed All Follow-up | 23 | 21 | 36
Included in Analysis (Intent-to-treat analysis was primary: Treatment completion defined as: attending 6/8 CBTH sessions; attending 9/12 CPT sessions) | 65 (41 - contributed >= 1 HIT-6 outcome 40 - contributed >= 1 PCL-5 outcomes 65 - included in multiple imputation) | 64 (27 - contributed >= 1 HIT-6 outcome 26 - contributed >= 1 PCL-5 outcomes 64 - included in multiple imputation) | 64 (51 - contributed >= 1 HIT-6 outcome 51 - contributed >= 1 PCL-5 outcomes 64 - included in multiple imputation)
Completed (Completed all sessions) | 33 | 23 | 48
Not Completed | 22 | 25 | 9
Not completed — Withdrawn or lost to follow-up | 22 | 25 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Headache Therapy | Cognitive Processing Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 65 | 64 | 64 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (8.4) | 39.7 (8.4) | 39.7 (8.4) | 39.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 individual did not report gender
  Participants
    number analyzed (Participants) | 65 | 64 | 63 | 192
    Female | 9 | 6 | 10 | 25
    Male | 56 | 58 | 53 | 167
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 2 individuals did not report ethnicity
  Participants
    Ethnicity: number analyzed (Participants) | 64 | 64 | 63 | 191
    Ethnicity: Hispanic | 27 | 28 | 26 | 81
    Ethnicity: Non-Hispanic | 37 | 36 | 37 | 110
Race [Count of Participants; unit: Participants] — Population: 2 individuals did not report race
  Participants
    number analyzed (Participants) | 65 | 63 | 63 | 191
    American Indian | 0 | 1 | 4 | 5
    Asian | 2 | 1 | 4 | 7
    Black/African American | 7 | 14 | 13 | 34
    Native Hawaiian | 2 | 2 | 2 | 6
    White | 43 | 34 | 33 | 110
    Other | 11 | 11 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Headache-related Disability Scores on the Headache Impact Test 6 (HIT-6)
Description: Baseline headache-related disability will be assessed over time based on headache-related disability scores on the HIT-6 obtained at multiple time points: at the end of 6 weeks of treatment, and at 3 and 6 months post-treatment. The Headache Impact Test (HIT-6) is a questionnaire for measuring the impact of headache. A total of six questions are completed by the patient. They focus on daily activities such as work, education, home situation and leisure time. The HIT-6 gives a general overview of the impact of headache, including pain intensity, impairment and other items. Each of the six questions of the HIT-6 receives a score from 6-13. The final HIT-6 score can range from 36 to 78. A higher score indicates more disability due to headache.
Time Frame: Baseline, 6 weeks (end of treatment), and 3 and 6 months post-treatment
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Behavioral Headache Therapy: A standard, manualized behavioral intervention for primary headache disorders
  Behavioral Headache Therapy: A standard, manualized behavioral intervention for primary headache disorders
  41 - contributed >= 1 HIT-6 outcome 40 - contributed >= 1 PCL-5 outcomes 65 - included in multiple imputation
Arm/Group | Behavioral Headache Therapy | Cognitive Processing Therapy | Treatment as Usual
Number analyzed (Participants) | 65 | 64 | 64
score on a scale
  Baseline | 66.1 (5.4) | 66.1 (5.1) | 65.2 (6.4)
  Post-treatment | 61.9 (6.3) | 63.3 (6.9) | 64.2 (6.6)
  3-Month Follow-up | 61.3 (8.0) | 64.8 (7.2) | 64.1 (7.1)
  6-Month Follow-up | 60.9 (8.8) | 63.3 (7.1) | 64.1 (7.3)
Statistical Analysis 1: Comparison: Behavioral Headache Therapy vs Cognitive Processing Therapy vs Treatment as Usual; Sample size based on 2-tailed specified joint superiority testing of 2 primary outcomes at α = .025 and power of 0.80 to detect an effect size (d) of 0.52 for both primary outcomes (representing a clinically significant change of 2.8 points on the HIT-6). The primary analysis set was intention to treat (ITT). multiple imputation accounted for missing data in ITT. Missing outcome scores at posttreatment, 3-month, and 6-month follow-ups were multiply imputed (m = 100) using multilevel models; Test type: Superiority — Superiority of the experimental arms (CBTH and CPT) compared to usual care (TAU); p < 0.001, Mixed Models Analysis — p-value represents an aggregate of post-treatment outcomes (i.e., post-treatment, 3-month, and 6-month outcomes entered simultaneously into the GLMM to represent a single metric of all post-treatment assessment intervals into one estimate); Outcome observations at posttreatment, 3-month and 6-month follow-ups were entered simultaneously into the mixed model to provide a single inference; Aggregated contrast CBTH to TAU = -3.4, 95% CI 2-sided [-5.4 to -1.4] — Contrast of aggregated post-treatment outcomes of HIT-6 total score for CBTH compared to TAU
Statistical Analysis 2: Comparison: Behavioral Headache Therapy vs Cognitive Processing Therapy vs Treatment as Usual; See previous section for power; Test type: Superiority — See previous section for analysis; p = 0.21, Mixed Models Analysis — For comparison of post-treatment HIT-6 total score between CPT and TAU; See above for details; Aggregated contrast CPT to TAU = -1.4, 95% CI 2-sided [-3.7 to 0.8] — See above

2. Primary Outcome: Scores for Symptoms of Post-traumatic Stress on the PTSD Checklist-5 (PCL-5)
Description: Post-traumatic stress scores will be assessed over time. The PTSD Checklist for DSM-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. Respondents are asked to rate how bothered they have been by each of 20 items in the past month on a 5- point. Likert scale ranging from 0-4. Items are summed to provide a total severity score (range = 0-80). A higher score indicates more PTSD.
  0 = Not at all 1 = A little bit 2 = Moderately 3 = Quite a bit 4 = Extremely
Time Frame: Baseline, 6 weeks (end of treatment), and 3 and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Headache Therapy | Cognitive Processing Therapy | Treatment as Usual
Number analyzed (Participants) | 65 | 64 | 64
score on a scale
  Baseline | 47.7 (14.7) | 48.6 (14.6) | 49.0 (13.3)
  Post-Treatment | 36.5 (19.7) | 30.0 (20.9) | 41.6 (17.1)
  3-Month Follow-up | 30.2 (18.2) | 29.9 (20.0) | 43.0 (16.5)
  6-Month Follow-up | 30.3 (20.0) | 32.9 (21.0) | 41.0 (16.1)
Statistical Analysis 1: Comparison: Behavioral Headache Therapy vs Cognitive Processing Therapy vs Treatment as Usual; Same sample size calculation as HIT-6 analyses, powered to detect a difference of 8.2 points on the PCL-5 total score; Test type: Superiority — Key parameters and details the same as HIT-6 described above; p = 0.04, Mixed Models Analysis — Contrast of aggregate post-treatment outcomes between CBTH and TAU; Contrast of aggregate post-treatment outcomes between CBTH and TAU; Aggregated contrast CBTH to TAU = -6.5, 95% CI 2-sided [-12.7 to -0.3]
Statistical Analysis 2: Comparison: Behavioral Headache Therapy vs Cognitive Processing Therapy vs Treatment as Usual; See above; Test type: Superiority — Contrast of aggregate post-treatment outcomes between CPT and TAU; p = 0.01, Mixed Models Analysis — Contrast of aggregate post-treatment outcomes between CPT and TAU; Contrast of aggregate post-treatment outcomes between CPT and TAU; Aggregated contrast CPT to TAU = -8.9, 95% CI 2-sided [-15.9 to -1.9]

ADVERSE EVENTS:
Time Frame: Baseline to 6-month post-treatment follow-up for a total of approximately 7 months (+/- 2 weeks).
Description: Adverse events were gathered at all study visits (i.e., treatment and assessment visits) and TAU participants were contacted twice during the treatment phase to assess for adverse events.
Arm/Group | Behavioral Headache Therapy | Cognitive Processing Therapy | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/65 | 2/64 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Headache Therapy (N=65) | Cognitive Processing Therapy (N=64) | Treatment as Usual (N=64)
Hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) — Suicidal risk
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Headache Therapy (N=65) | Cognitive Processing Therapy (N=64) | Treatment as Usual (N=64)
Worsening PTSD symptoms (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) — PCL-5 score increase

LIMITATIONS AND CAVEATS:
Trial limitations include the chosen primary outcome, blinding a behavioral trial, definition of PTH as headache onset within 3 months of head injury (instead of 7 days per ICHD-3 5.2.2), and missing data/dropout. Dropout and missing data from this trial were high, though consistent with dropout risk in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT02419131/Prot_SAP_000.pdf